CLINICAL TRIAL: NCT05055245
Title: Stress in Couples Undergoing Assisted Reproduction Technology With Different Cycles and Its Impact on Pregnancy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Principal Investigator, Yimin Zhu, Chief Physician, Women's Hospital School Of Medicine Zhejiang University
Other Study IDs: 20210914
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Infertility
Keywords: infertility; cycle
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing assisted reproductive technology: Patients undergoing in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI)
  Interventions: Other: cycles

INTERVENTIONS:
Other: cycles — Patients are grouped according to the number of IVF/ICSI cycles.

SUMMARY:
With the development of assisted reproductive technology (ART), more and more infertile women are obtaining their offspring through assisted reproductive technology. However, a growing number of national and international studies have shown that infertility patients are prone to negative emotions such as anxiety and depression during ART treatment, which not only affects their physical and mental health, but also affects the embryo implantation rate and pregnancy rate of ART. The purpose of this study is to investigate the stress faced by participants undergoing ART with different cycles and to further investigate its impact on pregnancy outcomes.

DETAILED DESCRIPTION:
With the rapid social and economic development in recent years, the incidence of infertility has increased significantly due to environmental pollution, poor lifestyle habits and increasing stress in various areas. According to global statistics, one in six married couples suffers from infertility. With the development of assisted reproductive technology (ART), more and more infertile women are obtaining their offspring. In clinical practice, however, a significant proportion of patients undergoing ART have low embryo implantation and pregnancy rates and experience recurrent implantation failure (RIF). A growing number of national and international studies have shown that infertility patients are prone to negative emotions such as anxiety and depression during ART treatment, which not only affects their physical and mental health, but also affects the embryo implantation rate and pregnancy rate of ART. This effect is more pronounced in patients with multiple failed transfers. In this study, investigators intend to investigate the stress faced by participants undergoing assisted reproduction with different cycles to provide a reliable basis for future psychological interventions and health education for this group of patients and improve the quality of life of infertility patients.

ELIGIBILITY:
Inclusion Criteria:

* Female partners' >18< 40 years
* Patients undergoing assisted reproductive technology

Exclusion Criteria:

* Female partners with polycystic ovary
* Female partners with insufficiency or premature ovarian failure
* Female partners with endometriosis
* Female partners with abnormal profile of thyroid hormones
* Chromosomal abnormalities of either spouse
* Mental disorder of either spouse

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients undergoing assisted reproductive technology
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-09 (Estimated); Primary Completion 2022-03-09 (Estimated); Study Completion 2022-04-09 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 6 months
  Implantation rate is defined as number of sacs per embryo transferred.
clinical pregnancy rate | 6 months
  presence of at least one gestational sac on ultrasound of 6 weeks

SECONDARY OUTCOMES:
fertilization rate | 6 months
  No. of fertilized oocyte divided by No. of inseminated cumulus-oocyte complexes (COCs)
cleavage rate | 6 months
  No. of cleaved embryo divided by No. of fertilized oocyte
Total gonadotropin use | 6 months
  Total gonadotropin use of each participant
Ovarian hyperstimulation syndrome (OHSS) rates | 6 months
  OHSS rates in both study groups
Number of oocytes retrieved | 6 months
Metaphase II (MII) oocytes | 6 months
  the number of mature oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Zhu, Dr., Study Chair — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China